CLINICAL TRIAL: NCT05583227
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Phase 3 Efficacy and Safety Study of Tezepelumab in Patients With Eosinophilic Esophagitis (CROSSING).
Brief Title: Efficacy and Safety of Tezepelumab in Patients With Eosinophilic Esophagitis
Acronym: CROSSING
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5244C00001; 2022-001294-31 (EudraCT Number)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: Chronic Esophagitis; Eosinophilic Esophagitis; Eosinophilic
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1:1 ratio to receive either low dose of tezepelumab, high dose of tezepelumab, or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tezepelumab Low Dose (Experimental): Tezepelumab subcutaneous injections, in accessorised pre-filled syringes
  Interventions: Biological: Tezepelumab
- Tezepelumab High Dose (Experimental): Tezepelumab subcutaneous injections, in accessorised pre-filled syringes
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Placebo subcutaneous injections, in accessorised pre-filled syringes
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab Low Dose
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab High Dose
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled multicenter, phase 3 study to evaluate the efficacy and safety of tezepelumab administered subcutaneously (SC) using an accessorized pre-filled syringe (APFS) versus placebo in adult and adolescent patients with eosinophilic esophagitis (EoE).

DETAILED DESCRIPTION:
The study consists of a screening period of 2 to 8 weeks and a 52-week randomized double-blind placebo-controlled treatment period. After completion of the treatment period, participants will be eligible to participate in an optional active treatment extension period (lasting for 24 weeks), followed by a 12-week off-treatment safety follow-up period. Participants who will not participate in the extension period will participate in a 12-week off-treatment safety follow-up period following completion of the 52-week treatment period.

This study will randomize approximately 360 participants. The participants will be randomized at 1:1:1 ratio to the 3 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 12 to 80 years of age inclusive, at the time of signing the informed consent/assent.
2. Weight ≥ 40 kg at Visit 1
3. Established diagnosis of EoE with a previous EGD and esophageal biopsy confirming a diagnosis of EoE.
4. Participants who have symptomatic EoE as defined by a history of on average at least 2 episodes of dysphagia (any severity of food going down slowly or being stuck in the throat) per week in the 4 weeks prior to Visit 1.
5. Must remain on a stabilized diet for at least 8 weeks prior to Visit 1 and during the course of the study (stable diet is defined as no initiation of single or multiple elimination diets or reintroduction of previously eliminated food groups).
6. May be on any background PPI and/or STC, during the course of the study, as long as background medications have been stable for at least 8 weeks prior to the screening/run-in period (Visit 1) and there is agreement not to change background medication or dosage unless medically indicated, during the screening/run-in and treatment period.
7. Participants currently on leukotriene inhibitors and/or steroid treatments for asthma or allergies that are inhaled or administered intranasally, must report a stable dose for at least 4 weeks prior to the screening/run-in period (Visit 1).
8. If a medication for EoE (for example PPI and/or STC) is discontinued prior to the screening/run-in, there should be a washout period of at least 8 weeks prior to Visit 1. Discontinuation of any marketed biologic (monoclonal or polyclonal antibody) should have a washout period of 4 months or 5 half-lives prior to Visit 1, whichever is longer.
9. Participants should have previously documented standard of care treatment, which could include PPI and/or STC and/or diet.

Exclusion Criteria:

1. Other gastrointestinal disorders such as active Helicobacter pylori infection, history of achalasia, esophageal varices, Crohn's disease, ulcerative colitis, inflammatory bowel disease, celiac disease, eosinophilic enteritis, colitis, diverticulitis, irritable bowel syndrome, or other clinically significant gastrointestinal conditions as per Investigator discretion.
2. Esophageal stricture that prevents the easy passage of a standard endoscope or any critical esophageal stricture that requires dilation at screening.
3. Use of a feeding tube, or having a pattern of not eating solid food >3 days of week. Solid food is defined as food that requires chewing before swallowing.
4. Hypereosinophilic syndrome
5. EGPA vasculitis
6. Esophageal dilation performed within 8 weeks prior to screening.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
Histologic response of peak esophageal eosinophil per HPF count of ≤ 6 across all available esophageal levels | Week 24
  Peak esophageal eosinophil count per HPF determined by histological analysis of 2-4 biopsies from each of the proximal, mid, and distal esophagus.
Change from baseline in DSQ (Dysphagia Symptom Questionnaire) score | Week 24
  The Dysphagia Symptom Questionnaire (DSQ) captures the presence and severity of dysphagia symptoms in the past day in a 4-item questionnaire. The DSQ score is calculated over 14-day periods and ranges from 0 to 84, with a lower score indicating less severe dysphagia.

SECONDARY OUTCOMES:
Change from baseline in EoE EREFS (Endoscopic reference score ) | Week 24, Week 52
  The EoE EREFS is a scoring system for assessing the presence and severity of the major endoscopic signs of EoE, including esophageal edema, rings, exudates, furrows, and stricture.
  EoE endoscopic appearances will be analyzed by the EoE-EREFS, a scoring system for inflammatory and fibrostenotic features of the disease. Proximal and distal esophageal areas will be scored, with the score for each region ranging from 0 to 9, and the overall score ranging from 0 to 18. Higher scores indicate more extensive disease.
Change from baseline in EoE-HSS (Histologic scoring system) grade score | Week 24
  EoE HSS is a histology scoring system for esophageal biopsies that evaluates 8 features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. Severity (grade) and extent (stage) of abnormalities are scored using a 4-point scale (0 normal; 3 maximum change).
Change from baseline in EoE-HSS (Histologic scoring system) stage score | Week 24
  EoE HSS is a histology scoring system for esophageal biopsies that evaluates 8 features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. Severity (grade) and extent (stage) of abnormalities are scored using a 4-point scale (0 normal; 3 maximum change).
Histologic response of peak esophageal eosinophil per HPF count of ≤ 6 across all available esophageal levels | Week 52
  The peak esophageal eosinophil count is based on 2-4 esophageal biopsies from 2-3 locations.
Change from baseline in DSQ (Dysphagia Symptom Questionnaire) score | Week 52
  The Dysphagia Symptom Questionnaire (DSQ) captures the presence and severity of dysphagia symptoms in the past day in a 4-item questionnaire. The DSQ score is calculated over 14-day periods and ranges from 0 to 84, with a lower score indicating less severe dysphagia.
Endoscopic response of total EREFS score of 0 to ≤2 with no score > 1 for any of the components and no worsening in any individual component from baseline accross all esophageal levels | Week 52
  EoE endoscopic appearances will be analyzed by the EoE-EREFS, a scoring system for inflammatory and fibrostenotic features of the disease. For each of the EREFS compontents a maximum score across proximal, mid and distal esophageal areas will be selected, with the scores for edema and stricture ranging from 0 to 1, exudates and furrows ranging from 0 to 2, fixed rings ranging from 0 to 3, and overall maximum score ranging from 0 to 9.
Endoscopic inflammatory remission of EREFS inflammatory subscore (including edema, exudate, and furrows components) of 0 with no worsening in rings or stricture from baseline across all esophageal levels) | Week 52
  EoE endoscopic appearances will be analyzed by the EoE-EREFS, a scoring system for inflammatory and fibrostenotic features of the disease. For each of the EREFS compontents a maximum score across proximal, mid and distal esophageal areas will be selected, with the scores for edema and stricture ranging from 0 to 1, exudates and furrows ranging from 0 to 2, fixed rings ranging from 0 to 3, and overall maximum score ranging from 0 to 9.
Total endoscopic remission of total EREFS score of 0 across all esophageal levels | Week 52
  EoE endoscopic appearances will be analyzed by the EoE-EREFS, a scoring system for inflammatory and fibrostenotic features of the disease. For each of the EREFS compontents a maximum score across proximal, mid and distal esophageal areas will be selected, with the scores for edema and stricture ranging from 0 to 1, exudates and furrows ranging from 0 to 2, fixed rings ranging from 0 to 3, and overall maximum score ranging from 0 to 9.

OTHER OUTCOMES:
Change from baseline in peak esophageal eosinophil count (EOS/HPF) | Week 24, Week 52
  The EOS/HPF is a method of evaluating esophageal inflammation by histological response of eosinophils per high power field (HPF).
Changes from baseline in PEESS Module at Week 24 (adolescents only). | Week 24, Week 52
  The PEESS is an 20-item assessment of EoE symptom severity and frequency validated for use in patients aged 8 to 18 years. The overall score ranges from 0 to 80, with higher scores representing more severe and frequent EoE symptoms.
Change from baseline in EoE-HSS (Histologic scoring system) stage score | Week 52
  EoE HSS is a histology scoring system for esophageal biopsies that evaluates 8 features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. Extent (stage) of abnormalities is scored using a 4-point scale (0 normal; 3 maximum change).
Change from baseline in EoE-HSS (Histologic scoring system) grade score | Week 52
  EoE HSS is a histology scoring system for esophageal biopsies that evaluates 8 features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. Severity (grade) of abnormalities is scored using a 4-point scale (0 normal; 3 maximum change).
Serum tezepelumab concentration | Weeks 0, 4, 12, 24, and 52
  PK samples will be collected pre-dose. Tezepelumab concentration in serum is determined using bioanalytical method.
Anti-drug antibody | Weeks 0, 12, 24, and 52
  Anti-drug antibody is determined using bioanalytical method.

CONTACTS AND LOCATIONS:
Locations (109):
- United States (23):
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Normal, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Chesterfield, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Ocean City, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
- Australia (4):
  - Research Site, Elizabeth Vale
  - Research Site, Kogarah
  - Research Site, South Brisbane
  - Research Site, Woolloongabba
- Austria (2):
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (4):
  - Research Site, Bruges
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Brazil (7):
  - Research Site, Botucatu
  - Research Site, Brasília
  - Research Site, Caxias do Sul
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
- China (8):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Køge
  - Research Site, Odense
- Research Site, Helsinki, Finland
- Research Site, München, Germany
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Israel (5):
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (8):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Verona
- Japan (12):
  - Research Site, Akita
  - Research Site, Fukuoka
  - Research Site, Himeji
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Maebashi
  - Research Site, Minatoku
  - Research Site, Osaka
  - Research Site, Shinjuku-ku
  - Research Site, Yamagata
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- New Zealand (4):
  - Research Site, Christchurch
  - Research Site, Hamilton
  - Research Site, Newtown
  - Research Site, Otahuhu
- Norway (4):
  - Research Site, Ålesund
  - Research Site, Lørenskog
  - Research Site, Oslo
  - Research Site, Tromsø
- Research Site, Košice, Slovakia
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Tomelloso
- Sweden (3):
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Uppsala
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: This webpage was designed to learn about the work AstraZeneca is doing to develop Eosinophilic Esophagitis (EoE) treatments and find out how you could get involved in a clinical trial. — https://www.eoetrialandyou.com/en-US/selector/all